CLINICAL TRIAL: NCT06383845
Title: Comparison of Erector Spinae Plane Block and Intravenous Lidocaine for Chronic Pain Post Mastectomy: a Randomized Controlled Trial
Brief Title: Comparison of Erector Spinae Plane Block vs Intravenous Lidocaine for Chronic Pain Post Mastectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, HibetAllah Ktata, Associate Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MAS ESLI
Record Dates: First submitted 2024-04-14; First posted 2024-04-25 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Surgery

STUDY DESIGN:
Intervention Model Description: Erector spinae plane block VS intravenous lidocaine.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine-IV (Experimental): Intravenous Lidocaine dose loading than continuous infusion
  Interventions: Drug: Lido-IV
- Erector spinae Block (Active Comparator): An ultrasound guided Erector Spinae Block is performed with injection of 30 ml of Ropivacaine 3.75%
  Interventions: Drug: ESP Block

INTERVENTIONS:
Drug: Lido-IV — Intravenous Lidocaine dose loading than a continuous infusion
  Other Names: Lidocaine-IV
  Arms: Lidocaine-IV
Drug: ESP Block — ultrasound guided block with injection of Ropivacaine
  Other Names: Erector Spinae Block
  Arms: Erector spinae Block

SUMMARY:
Patients undergoing breast surgery were divided into two groups: Intravenous Lidocaine (Lido-IV) vs Erector Spinae Block (ESP).

For Lido-IV group, patients received a loading dose of Lidocaine than a continuous infusion till the end of surgery.

For ESP group, an ultrasound guided ESP Block was perormed before anesthetic induction.

Persistant pain post mastectomy was assessed by SFM-PQ score at 1, 3 and 6 months post surgery.

DETAILED DESCRIPTION:
Patients undergoing breast surgery with lymph node dissection were divided into two groups: Intravenous Lidocaine (Lido-IV) vs Erector Spinae Block (ESP).

For Lido-IV group, patients received a loading dose of 1.5 mg/kg of Lidocaine than a continuous infusion of 2 mg/kg/h till the end of surgery.

For ESP group, an ultrasound guided ESP Block was perormed before anesthetic induction with injection of 30 ml of Ropivacaine 3.75%.

For both group, persistant pain post mastectomy was assessed by Item 5 of BPI score at 1, 3 and 6 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* patients aged 18 and older
* American Society of anesthesiologists classification I or II
* patients proposed for planned mastectomy with axillary lymph node dissection.
* hemodynamic stability.

Exclusion Criteria:

* patient refusal
* male gender
* history of major surgery within the year.
* allergy to local anesthetics
* BMI>40
* hemodynamic instability
* Patients on long-term analgesics
* Severe heart and/or kidney damage
* neurological/psychiatric impairment

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Item 5 of Brief Pain inventory score (BPI Score) | item 5 of the BPI score evaluated as follows: 0 minimum score and 10 maximum score, at 01, 03 and 06 months post surgery
  Note of Brief Pain inventory Scale (BPI Score)

SECONDARY OUTCOMES:
Acute pain assessed by Simple Verbal Scale (SVS) | Postoperatively, at Hour 2, Hour 12 and Hour 24
  Acute Postoperative pain was assessed by the Simple Verbal Scale (SVS)
Postoperative nausea and vomiting | During the first 24hours postoperatively
  Incidence of postoperative nausea and vomiting during the first 24 hours
Hospital length of stay | From the end of the surgery to discharge from the hospital
  hospital length of stay (in days)
DN4 questionnaire (DN4) | DN4 represented by 10 items with a score from a minimum of 0 to a maximum of 10, at 03 and 06 months post surgery
  DN4 questionnaire scale
The short-form McGill Pain Questionnaire (SFM-PQ) | the 15 items are rated on a four-point pain intensity scale, at 01, 03 and 06 months after surgery
  The short-form McGill Pain Questionnaire Scale: Sensory and affective components of pain (11 sensory items and 4 affective items)

CONTACTS AND LOCATIONS:
Locations (1):
- Tunisia, Nabeul, Tunisia